CLINICAL TRIAL: NCT01733108
Title: An Open-Label Drug-Drug Interaction Study in Healthy Subjects to Explore the Effects of Multiple Doses of JNJ-28431754 on the Pharmacokinetics and Safety of Single Doses of Glyburide
Brief Title: A Study to Assess the Effects of Canagliflozin (JNJ-28431754) on the Pharmacokinetics, Pharmacodynamics, and Safety of Glyburide in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014872; 28431754DIA1004 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C)
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Healthy; Canagliflozin (JNJ-28431754); Pharmacokinetics; Pharmacodynamics; Glyburide (MICRONASE)
MeSH Terms: interventions — Glyburide; Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Canagliflozin (JNJ-28431754) + glyburide (Experimental): Each volunteer will receive a single dose of glyburide on Day 1, followed by canagliflozin (JNJ-28431754) once daily on Days 4 through 8. On Day 9 volunteers will receive a single dose of glyburide in combination with a single dose of canagliflozin.
  Interventions: Drug: Glyburide; Drug: Canagliflozin (JNJ-28431754)

INTERVENTIONS:
Drug: Glyburide — One 1.25 mg tablet taken orally (by mouth) on Day 1 and Day 9.
  Other Names: Micronase
Drug: Canagliflozin (JNJ-28431754) — One 200 mg tablet taken orally (by mouth) on Days 4 through 9.
  Other Names: JNJ-28431754

SUMMARY:
The purpose of this study is to determine how multiple doses of canagliflozin (JNJ-28431754) affect the pharmacokinetics (ie, how the body affects the drug) and pharmacodynamics (ie, how the drug affects the body) of a single dose of glyburide.

DETAILED DESCRIPTION:
This study will be an open-label (all volunteers and study staff know the identity of the assigned treatment), single-center, fixed-sequence study (all volunteers receive the same medication on the same days) to determine how canagliflozin (a drug currently being investigated for the treatment of type 2 diabetes mellitus) affects the pharmacokinetics and pharmacodynamics of glyburide (a blood glucose-lowering agent used to treat patients with diabetes). The study will consist of 3 phases; a screening phase, an open-label treatment phase, and an end-of-study (or follow-up) phase. During the open-label treatment phase, each volunteer will receive a single 1.25 mg dose of glyburide on Day 1, followed by 200 mg canagliflozin once daily on Days 4 through 8. On Day 9 volunteers will receive both glyburide 1.25 mg and canagliflozin 200 mg. Each volunteer will participate in the study for approximately 40 days.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer must have a body mass index (BMI = weight in kg/height in m2) between 18 and 30 kg/m2 (inclusive) and body weight not less than 50 kg Exclusion Criteria:
* Volunteer has a history of or currently active illness considered to be clinically significant by the Investigator or any other illness that the Investigator considers should exclude the patient from the study or that could interfere with the interpretation of the study results
* Volunteer has a fasting plasma glucose < 100 mg/dL (as measured by oral glucose tolerance test) and a 2-hour plasma glucose <= 140 mg/dL
* History of smoking or use of nicotine-containing substances within the previous 6 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of glyburide | Up to Day 12
  Comparison of plasma concentrations of glyburide following administration of a single dose of glyburide alone or in combination with multiple doses of canagliflozin (JNJ-28431754). This will be used to determine whether there is a pharmacokinetic interaction between glyburide and canagliflozin.
Plasma concentrations of glyburide metabolites | Up to Day 12
  Comparison of plasma concentrations of glyburide metabolites following administration of a single dose of glyburide alone or in combination with multiple doses of canagliflozin (JNJ-28431754). This will be used to determine whether there is a pharmacokinetic interaction between glyburide and canagliflozin.

SECONDARY OUTCOMES:
Change from baseline in plasma glucose concentrations | Day -1 (Baseline) up to Day 9
  Plasma glucose concentrations following the administration of a single dose of glyburide after the administration of multiple doses of canagliflozin (JNJ-28431754) will be used to determine whether there is a pharmacodynamic interaction (changes in plasma glucose) between glyburide and canagliflozin. The area under the plasma glucose concentration-time curve (AUC) will be used as the key pharmacodynamic parameter.
Change from baseline in plasma insulin concentrations | Day -1 (Baseline) up to Day 9
  Plasma insulin concentrations following the administration of a single dose of glyburide after the administration of multiple doses of canagliflozin (JNJ-28431754) will be used to determine whether there is a pharmacodynamic interaction (changes to plasma insulin) between glyburide and canagliflozin. The area under the plasma insulin concentration-time curve (AUC) will be used as the key pharmacodynamic parameter.
Change from baseline in plasma C-peptide concentrations | Day -1 (Baseline) up to Day 9
  Plasma C-peptide is formed during the body's production of insulin. Plasma C-peptide concentrations following the administration of a single dose of glyburide after the administration of multiple doses of canagliflozin (JNJ-28431754) will be used to determine whether there is a pharmacodynamic interaction (changes to plasma C-peptide) between glyburide and canaglifloxin. The area under the plasma C-peptide concentration-time curve (AUC) will be used as the key pharmacodynamic parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Devineni D, Manitpisitkul P, Murphy J, Skee D, Wajs E, Mamidi RN, Tian H, Vandebosch A, Wang SS, Verhaeghe T, Stieltjes H, Usiskin K. Effect of canagliflozin on the pharmacokinetics of glyburide, metformin, and simvastatin in healthy participants. Clin Pharmacol Drug Dev. 2015 May-Jun;4(3):226-36. doi: 10.1002/cpdd.166. Epub 2014 Oct 27. PMID 27140803